CLINICAL TRIAL: NCT06501560
Title: Profiles Analysis of Genome Wide Association Study (GWAS) in Acne Vulgaris in Indonesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Collaborators: Indonesia Medical Education and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. Dr. dr. Irma Bernadette S. Sitohang, Sp.KK (K), Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Univ_Indo
Record Dates: First submitted 2024-06-02; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Acne Vulgaris
Keywords: Acne; Acne Vulgaris (AV); Genome Wide Association Study (GWAS); Genetic; Genotype; Deoxyribonucleic Acid (DNA); Single Nucleotide Polymorphism (SNP)
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle counseling (Experimental)
  Interventions: Genetic: GWAS
- clinical examination (Experimental)
  Interventions: Genetic: GWAS

INTERVENTIONS:
Genetic: GWAS — In GWAS studies, data are collected to determine common variants in a number of individuals, either with or without a common trait (for example,. disease) across the genome, using genome wide SNP arrays.

SUMMARY:
This study is a series of descriptive-analytic studies on genomic variants in the facial skin of patients with AV at the Dermatology and Venereology Polyclinic by determining the genetic profile by GWAS examination in AVB and analysing the genetic profile in AVB against differences in geographical location. The research design used was a cross-sectional design.

DETAILED DESCRIPTION:
Research subjects were obtained from the affordable population who met the research criteria and expressed their willingness to participate in the study.

Subject selection was carried out by purposive sampling method that met the inclusion criteria. The study will be conducted in one visit where the patient and his/her parents come to be given an explanation about the study with a request for informed consent, screening for inclusion and exclusion criteria, anamnesis of facial complaints, taking data on demographics, patient's medical history, patient's medical history, physical examination, taking clinical photos in 5 positions and ending with taking blood samples of the patient and blood samples from both parents of the patient as much as 10 mL.

The study will be conducted in three places, namely in Jakarta, Padang, and Manado. In sampling in Padang and Manado, to prevent damage to the samples that have been taken, the samples will be stored at a temperature of -20C, then when brought to Jakarta will use a cooler box along with an ice pack at a temperature of 2-3C, before being processed in the Bioinformatics Core Facilities IMERI laboratory, Jakarta. When the samples are collected in Jakarta, the blood samples will be immediately stored in the laboratory at -20C.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with AVB aged 17-21 years
* Both parents of complete subjects with or without a history of acne vulgaris aged up to 60 years
* Patients and parents are willing to participate in the study and sign informed consent.

Exclusion Criteria:

* Patients who have other inflammatory or infectious diseases especially on the face
* Have genetic diseases or disorders
* Diagnosed with primary or secondary immunodeficiency diseases
* Using oral or systemic antibiotic, anti-inflammatory, retinoid or hormone therapy in the past month.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
Severity of acne vulgaris | 1 year
  Physical examination: identify the number of blackheads, papules, pustules and cysts.
  Degree of severity:(1)Mild =Comedo<20, or inflammatory lesion<15, or total lesion<30(2)Moderate = Comedo 20-100, or inflammatory lesion15-50, or total lesion 30-125(3)Severe =cyst>5, or Comedo>100, or inflammatory lesion>50, or total lesion>125.
Population structure | 3 months
  Gene testing of blood sample Genetic Inflation Factor (GIF) >1.1 or <1.1 Principal Component Analysis (PCA)
Genomic Profile | 3 months
  Blood sample examination, processed using GWAS Mutations (SNPs)(1)Present(2)Absent
Linkage disequilibirium (LD) | 3 months
  Gene testing of blood samples Coefficient 0-1
Haplotype | 3 months
  Gene testing of blood samples Jumlah gen
  1. Satu gen
  2. Multipel gen
SNP Enrichment | 3 months
  Gene testing of blood samples Mutation position
Association analysis and Association analysis of imputation results | 3 months
  Gene testing of blood samples PCA value

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
The results of this study are expected to be the initial stage for further research on genetic profiles in AVB, Benefits for the Field of Community Service-Improve clinician knowledge about genetic profiles in AVB-The results of this study are expected to be used as a reference in acne vulgaris management services so that they can produce more measurable and effective therapy. and provide a positive impact for RSCM to improve optimal service to Dermatology and Venereology patients.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year
Access Criteria: data collection